CLINICAL TRIAL: NCT03315741
Title: The Safety and Tolerability of Pirfenidone for Bronchiolitis Obliterans Syndrome After Hematopoietic Cell Transplantation
Brief Title: The Safety and Tolerability of Pirfenidone for BOS After HCT
Acronym: STOP-BOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-43319; VAR0158 (Other: OnCore)
Record Dates: First submitted 2017-10-05; First posted 2017-10-20 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Bronchiolitis Obliterans; Graft Vs Host Disease
Keywords: Bronchiolitis obliterans syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans; Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: This is a phase 1, non-randomized, single arm, open label, single center clinical trial to determine the tolerability and safety of pirfenidone in patients with BOS associated with lung GVHD after hematopoietic cell transplant (HCT). Approximately 30 patients will be enrolled. All patients will follow the 'patient-centered' drug titration approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient centered approach (Experimental): Drug titration of maximum dose over 3-8 weeks
  Interventions: Drug: Pirfenidone 267 MG [Esbriet]

INTERVENTIONS:
Drug: Pirfenidone 267 MG [Esbriet] — Tolerability of drug

SUMMARY:
This is a phase 1, non-randomized, single-arm, open label, single center clinical trial to determine the tolerability and safety of pirfenidone in patients with BOS associated with lung GVHD after hematopoietic cell transplant.

DETAILED DESCRIPTION:
This is a phase 1, non-randomized, single-arm, open label, single center clinical trial to determine the tolerability and safety of pirfenidone in patients with BOS associated with lung GVHD after hematopoietic cell transplant (HCT). Such a trial is a necessary step prior to an evaluation of efficacy, as pirfenidone is known to be associated with adverse events (AEs) of the liver, gastrointestinal system and skin, organs frequently affected in GVHD. Approximately 30 patients will be enrolled, all patients will follow the same drug titration approach. The primary endpoint will be drug tolerability as measured by: the number of patients that are able to maintain the recommended dose of pirfenidone (2403 mg/d) without dose reduction lasting more than 21 days, due to adverse events (AEs). Changes from Baseline to Week 52 will be studied using validated health-related quality of life scales. Eligible patients aged > 18 years must have a diagnosis of BOS according to pre-specified criteria. Patients will be required to have an %FEV1 or %FVC decline >20% from pre-transplant baseline and symptoms of dyspnea, or cough. Eligible patients will enter the Screening Period, which may last up to 28 days. The dose of pirfenidone will be titrated over 3-8 weeks. Patients will have a telephone assessment at Week 1 and 2. An in-clinic assessment will occur every 1-3 months as part of their usual clinical care in the Stanford University Lung GVHD clinic. Patients will complete an AE and dosing compliance diary. If patients discontinue study treatment early for any reason, they will continue with all scheduled study procedures through Week 52. All deaths will be reviewed by a Mortality Assessment Committee (MAC). An external Data Safety Monitoring Board (DSMB) will monitor patient safety during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years at randomization
2. Clinical symptoms (e.g., dyspnea or cough) consistent with BOS of ≥ 2 months duration
3. Presence of cGVHD in an organ other than lung
4. Subjects must have had recent pulmonary function test (PFTs) measured for at least 3 months prior to study enrollment that show:

   1. A decrease in %FVC and/or %FEV1 ≥ 20% at Screening compared with pre-transplant baseline.
   2. Bronchodilator response on PFT testing that results in an FEV1 < 75%
5. Diagnosis of BOS by one of the following criteria:

   1. Transbronchial or surgical lung biopsy demonstrating the obliterative bronchiolitis lesion
   2. Volumetric CT scan with lung density analysis with ≥ 28% air trapping (1).
   3. NIH-based PFT criteria for the diagnosis of BOS: FEV1/FVC <0.7 and FEV1 < 75%
   4. Evidence of clinical improvement after treatment for BOS has been initiated.
6. No features supporting an alternative diagnosis by transbronchial biopsy, bronchoalveolar lavage (BAL), surgical lung biopsy, culture and non-culture based data, if performed
7. Adequate organ and marrow function including: liver function as defined by a total bilirubin below the upper limit of normal (ULN), excluding patients with Gilbert's syndrome; AST/SGOT or ALT/SGPT < 3 x ULN; alkaline phosphatase < 2.5 x ULN; renal function as defined by a CrCl > 30 mL/min, calculated using the Cockcroft-Gault formula; cardiac electrophysiologic stability as defined by an electrocardiogram (ECG) with a QTc interval < 500 msec at Screening; and bone marrow function as defined by a white blood cell count > 3 K/µL, an absolute neutrophil count > 15 K/µL and a platelet count > 20 K/µL
8. Life expectancy > 6 months
9. Participants must be able to understand and sign a written informed consent form and understand the importance of adherence to study treatment and protocol. In addition, participants must demonstrate a willingness to follow all study requirements, including the concomitant medication restrictions, throughout the study

Exclusion Criteria:

1. Any condition that, in the opinion of the investigator, might be significantly exacerbated by the known side effects associated with the administration of pirfenidone e.g., presence of active GVHD of the gastrointestinal tract as manifested by rising liver function tests (LFTs) prior to initiation of study treatment
2. Uncontrolled infection
3. Major surgery within the past 2 months
4. The use of another investigational drug within the previous 30 days.
5. Inability to attend scheduled clinic visits
6. Inability to perform pulmonary function testing
7. Significant clinical change in health in the past 30 days
8. Body mass index (BMI) < 17.5
9. Life expectancy < 6 months due to any condition other than BOS that, in the opinion of the investigator, is likely to result in the death of the patient.
10. History of unstable or deteriorating cardiac or pulmonary disease (other than BOS) within the previous 6 months, including but not limited to the following:

    1. Unstable angina pectoris or myocardial infarction
    2. Congestive heart failure requiring hospitalization
    3. Uncontrolled clinically significant arrhythmias
11. Pregnancy or lactation.
12. Family or personal history of long QT syndrome
13. Investigational therapy, defined as any drug that has not been approved for marketing for any indication in cGVHD will be restricted from the study
14. The following medications may significantly increase the level of Pirfenidone and should not be taken concurrently including: fluvoxamine, ciprofloxacin > 500mg twice daily, systemically administered aminolevulinic acid, vemurafenib and enoxacin. Any other strong inhibitors of P450 isoenzymes CYP1A2, CYP2C9, 2C19, 2D6, and 2E1 should be avoided. Participants that cannot take alternative medications to those listed above will be excluded from this study.

Laboratory Exclusions

1. Any of the following LFT criteria above specified limits: total bilirubin above the upper limit of normal (ULN), excluding patients with Gilbert's syndrome; aspartate or alanine aminotransferase (AST/SGOT or ALT/SGPT) >3 × ULN; alkaline phosphatase >2.5 × ULN
2. Creatinine clearance (CrCl) <30 mL/min, calculated using the Cockcroft-Gault formula
3. Electrocardiogram (ECG) with a QTc interval >500 msec at Screening

Medication Exclusions

1. Prior use of pirfenidone or known hypersensitivity to any of the components of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
The number of participants that do not require a reduction in drug dose for more than 21 days due to adverse events. | 52 weeks
  We will count the number of participants that do not require a reduction in drug dose of more than 21, non-continuous days due to adverse events. Tolerability will be assessed during continuous treatment. If the medication dosage increase results in the reoccurrence of a moderate adverse event or serious adverse event, lasting more than 21 days, then the event would be defined as "not tolerated". If adverse events resolve before 21 days, then participants will attempt to again up-titrate the Pirfenidone dose, as tolerated. If at least 25% of participants tolerate the drug, then investigators will deem that this study demonstrates adequate tolerability to proceed to a larger trial to examine drug efficacy.

SECONDARY OUTCOMES:
The number of participants that permanently discontinue drug due to adverse events. | 52 weeks
  We will count the number of patients that permanently discontinue Pirfenidone due to adverse events. A permanent discontinuation of drug is defined as discontinuation of the drug for more than 42 days.
The number of participants that temporarily discontinue drug due to adverse events. | 52 week
  We will count the number of participants that temporarily discontinue Pirfenidone due to adverse events. A temporary discontinuation of drug is defined as discontinuation of the drug for less than or equal to 42 days.
The number of patients that experience treatment-emergent adverse events | 56 week
  Treatment emergent events are defined as those that start or worsen after the start of study treatment and up to 28 days after the last dose of study treatment. AEs will be summarized by treatment group, system organ class, and preferred term, and also by the event's relationship to study treatment. At each level of summation, patients will be counted only once, under the greatest severity and strongest study-drug relationship (as reported by the investigator).
The number of patients that experience treatment-emergent serious adverse events (SAEs) | 56 week
  Serious adverse events (SAEs) are defined as those that result in: (i) death or are life threatening; (ii) result in hospitalization or prolong hospitalization; or (iii) result in disability (disruption of the participant's ability to conduct normal daily activities). Serious adverse events will be summarized by treatment group, system organ class, and preferred term, and also by the event's relationship to study treatment. At each level of summation, patients will be counted only once, under the greatest severity and strongest study-drug relationship (as reported by the investigator).
The number of patients that experience treatment-emergent deaths during the study period and for 28 days after the last dose of study treatment. | 56 week
  Treatment emergent deaths are defined as those that occur after the start of study treatment and up to 28 days after the last dose of study treatment and are deemed by the investigator to be related to study treatment.
All-cause mortality | 56 week
  We will count the total number of deaths during the study period and for 28 days after the last dose of study treatment
The number of patients that experience treatment-emergent changes in complete blood counts. | 52 week
  The complete blood count measures the number white blood cells (WBCs) per liter (L) including differential counts of the type of WBCs, hemoglobin concentration (g/dL), and platelet count per liter.
The number of patients that experience treatment-emergent changes in liver function testing. | 52 week
  We will assess treatment related changes in total bilirubin (mg/dL), AST/SGOT (units/L) or ALT/SGPT (units/L), alkaline phosphatase (units/L)
The number of patients that experience treatment-emergent changes in serum chemistries panel. | 52 week
  We will assess treatment related changes in potassium (mEq/L), blood urea nitrogen (mg/dL) and serum creatinine (mg/dL).
The number of patients that experience treatment-emergent changes in the corrected QT-interval on electrocardiogram. | 52 week
  We will evaluate changes in the interval from ventricular depolarization (Q-wave) to ventricular repolarization (T-wave) corrected for by heart rate
Body mass index | 52 week
  We will measure changes in the participant's height (meters) and weight (kg) to determine changes in body mass index (kg/m^2)
Oxygen saturation | 52 week
  We will measure the participant's oxygen saturation (%) at rest on room air.
Heart rate | 52 week
  We will measure the participant's resting heart rate (beats per minute)
Chronic GVHD assessment | 56 week
  Chronic GVHD symptoms will be assessed according to NIH cGVHD global severity score. The global cGVHD severity score evaluates the severity of cGVHD in eight sites including the skin, mouth, eyes, gastrointestinal track, liver, lungs, joints and fascia, and genital track. Each organ is assigned a severity score and composite scores are calculated based on the number of organs involved and the severity score within each affected organ.

OTHER OUTCOMES:
Pulmonary function testing: spirometric change from baseline to week 52. | 52 week
  We will measure the participant's Forced Expiratory Volume in 1 second (FEV1: L, % predicted), and Forced Vital Capacity (FVC: L, % predicted)
Pulmonary function testing: diffusion capacity for carbon monoxide (DLCO) change from baseline to week 52. | 52 week
  We will measure DLCO (ml/min/mmHg)
Change from Baseline to Week 52 in % air trapping as measured by volumetric CT thorax with lung density analysis | 52 week
  We will use lung density analysis to radiographically quantify the percent air trapping between an inspiratory and expiratory CT scan.
BOS-related mortality | 52 week
  We will count the number of participant deaths that are attributable to BOS.
Change from Baseline to Week 24 and 52 in dyspnea, as measured by the University of California at San Diego Shortness-of-Breath Questionnaire (UCSD SOBQ) score | 24 and 52 week
  Changes in dyspnea, as measured by UCSD SOBQ score, from Baseline to Week 26 and 52 will be analyzed using the same methods described in Section 5.4.2.1. Baseline UCSD SOBQ score will be the average of the measurements recorded at the Screening and Day 1 visits. The UCSD SOBQ score will be repeated at Week 26 and 52. The magnitude of the treatment effect of pirfenidone will be presented as the distribution (number and percentage) of patients across two categories of change from Baseline:
  * Increase of ≥ 25 points in the UCSD SOBQ score at Week 26 and 52 or death before Week 52
  * Decrease of ≥ 0
Change from Baseline to Week 24 and 52 in Chronic GVHD (cGVHD) response | 24 and 52 week
  The Lee cGVHD symptom scale contains 30 items in 7 subscales (skin, eye, mouth, lung, nutrition, energy and psychological), using a 5-point Likert scale. Scores are linearly transformed to a 0-100 scale with higher values representing more severe symptoms. A summary score also is calculated if 4 or more subscales are available for scoring. Change in GVHD symptoms as measured by the Lee GVHD-symptom scale from Baseline to Week 26 and 52 will be evaluated.
Cumulative systemic corticosteroid exposure | 52 week
  We will calculate the cumulative Prednisone dose (mg, or its corticosteroid equivalent) used by each participant over the trial period.
Use of other immunosuppressive medications | 52 week
  We will calculate the type and the cumulative dose (mg) of other immune suppressive medications used by each participant over the trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Joe L Hsu, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharifi H, Moss CT, Musa Z, Bell A, O'Donnell C, Borges CH, Matthaiou EI, Johnston L, Galban CJ, Sheshadri A, Yanik G, Cheng GS, Hsu JL. Pirfenidone for the treatment of bronchiolitis obliterans syndrome related to chronic graft-versus-host disease. Blood Adv. 2025 Oct 14;9(19):5024-5037. doi: 10.1182/bloodadvances.2025016122. PMID 40554417
- [Derived] Matthaiou EI, Sharifi H, O'Donnell C, Chiu W, Owyang C, Chatterjee P, Turk I, Johnston L, Brondstetter T, Morris K, Cheng GS, Hsu JL. The safety and tolerability of pirfenidone for bronchiolitis obliterans syndrome after hematopoietic cell transplant (STOP-BOS) trial. Bone Marrow Transplant. 2022 Aug;57(8):1319-1326. doi: 10.1038/s41409-022-01716-4. Epub 2022 May 31. PMID 35641662